CLINICAL TRIAL: NCT03320018
Title: Pilot Study of the Neuroprotective Effects of Hydrogen and Minocycline in Acute Ischemic Stroke
Brief Title: Neuroprotection in Acute Ischemic Stroke
Acronym: H2M
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Kamil Stefanowski, Clinical Assistant Professor of Neurology, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 932805
Record Dates: First submitted 2017-10-20; First posted 2017-10-24 (Actual); Results first posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Stroke, Ischemic
Keywords: neuroprotection; antioxidant
MeSH Terms: conditions — Ischemic Stroke | interventions — Hydrogen; Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hydrogen/Minocycline (Experimental): Hydrogen will be infused into aqueous solution (normal saline or water) at as high a concentration as possible (saturation = 1.6 ppm), and administered intravenously or orally respectively, TID for 3 days.
  Similarly, Minocycline will be administered either i.v. or p.o. once daily for 5 days.
  Interventions: Drug: Hydrogen; Drug: Minocycline
- Placebo Hydrogen/Placebo Minocycline (Placebo Comparator): Normal saline will be substituted for both Hydrogen and Minocycline for intravenous administration. Water will be substituted for hydrogen when administered p.o., and placebo capsules will be substituted for minocycline.
  Interventions: Other: Placebo Hydrogen; Other: Placebo Minocycline

INTERVENTIONS:
Drug: Hydrogen — Hydrogen will be infused into bags of normal saline solution and administered intravenously, or hydrogen generating tablets will be dissolved into water for the patient to drink, as the patient's condition permits. This will be administered TID for 3 days.
  Other Names: H2
  Arms: Hydrogen/Minocycline
Drug: Minocycline — Minocycline 200 mg will be mixed with normal saline and given by i.v. administration, or provided as capsules for the patient to swallow, q 24 hours for 5 days.
  Once patients regain the ability to swallow capsules, minocycline will be given orally in capsule form (2 capsules of 100 mg each), administered once daily for the remainder of the 5 day period.
  Other Names: Minocin; Minomycin; Akamin
  Arms: Hydrogen/Minocycline
Other: Placebo Hydrogen — Normal saline solution will be administered intravenously, in place of hydrogen solution.
  Placebo tablets will be dissolved into water for the patient to drink, as the patient's condition permits. This will be administered TID for 3 days.
  Arms: Placebo Hydrogen/Placebo Minocycline
Other: Placebo Minocycline — Normal saline solution or placebo capsule will be administered i.v. or p.o. respectively, in place of minocycline.
  Arms: Placebo Hydrogen/Placebo Minocycline

SUMMARY:
This is a pilot randomized control trial (RCT) to explore the possible beneficial effect of a novel combination therapy consisting of molecular hydrogen H2 plus minocycline ("H2M"), on neurological recovery after acute ischemic stroke.

DETAILED DESCRIPTION:
This will be a pilot trial exploring the ability of a novel combination ("H2M") of molecular hydrogen (an antioxidant) and minocycline (a widely used antibiotic known to inhibit the activation of matrix metallo-proteinase-9 and poly(ADP-ribose) polymerase), to protect brain tissue from ischemia/reperfusion injury that occurs during and after an ischemic stroke. Both hydrogen and minocycline have excellent safety profiles, have been previously demonstrated individually to reduce infarction in animal models of stroke, and have potentially synergistic mechanisms of action against ischemic brain damage. The mechanisms of action of both agents would be specifically relevant to patients receiving tissue plasminogen activator (tPA) or thrombectomy, and achieving some degree of therapeutic reperfusion.

This will be a double blinded, placebo-controlled trial. Eligible and willing subjects will be randomly assigned to be treated with either H2M or placebo, in addition to standard treatments. The treatment with H2M or placebo will start as soon as possible after diagnosis of stroke, and continue for three days (hydrogen) and five days (minocycline) respectively. Measures of stroke severity and disability will be recorded at baseline, and through a follow-up phone call (45 days) and clinic visit (90 days).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years old or over
2. Presenting to/at Stony Brook University Hospital with acute ischemic stroke
3. Baseline (at admission to study) National Institute of Health Stroke Scale (NIHSS) of ≥ 5
4. Administration of study medication possible within 24 hours of last known well

Exclusion Criteria:

1. Pre-existing neurological disability (historical NIHSS > 3); unable to live independently 3. Severe stroke or comorbidities likely to result in patient dying within 3 months 4. Acute or chronic renal failure with calculated creatinine clearance < 30 5. Liver disease leading to > 3x elevation in liver transaminases or significant loss of synthetic capacity* 6. Thrombocytopenia (<100x10^9platelets / L blood) 7. Pre-existing infectious disease requiring antibiotic therapy that have a negative interaction with minocycline. (Penicillin, amoxicillin, ampicillin, bacampicillin, carbenicillin, cloxacillin, dicloxacillin, methicillin, mezlocillin, nafcillin, oxacillin, piperacillin, ticarcillin) 8. Pregnancy or nursing. Females of reproductive age will be required to use barrier contraception or abstain from sexual intercourse while on study medications, as minocycline may render oral contraceptives less effective.

9. Known allergy to tetracycline group of drugs 10. Concurrent treatment with retinoids or ergot alkaloids 11. Inability to safely tolerate the fluid load (iv normal saline or po water) associated with study medication* 12. Treatment with another investigational drug within the last 30 days that may interfere with this study's medications* 13. Inability to tolerate or comply with study procedures*

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Choi, MD, PhD, Study Director — Stony Brook University Hospital
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 15 enrolled participants, 14 met inclusion exclusion criteria and were randomized to treatment.
Groups:
- Hydrogen/Minocycline: Hydrogen will be infused into aqueous solution (normal saline or water) at as high a concentration as possible (saturation = 1.6 ppm), and administered intravenously or orally respectively, TID for 3 days.
  Similarly, Minocycline will be administered either i.v. or p.o. once daily for 5 days.
  Hydrogen: Hydrogen will be infused into bags of normal saline solution and administered intravenously, or hydrogen generating tablets will be dissolved into water for the patient to drink, as the patient's condition permits. This will be administered TID for 3 days.
  Minocycline: Minocycline 200 mg will be mixed with normal saline and given by i.v. administration, or provided as capsules for the patient to swallow, q 24 hours for 5 days.
  Once patients regain the ability to swallow capsules, minocycline will be given orally in capsule form (2 capsules of 100 mg each), administered once daily for the remainder of the 5 day period.
- Placebo Hydrogen/Placebo Minocycline: Normal saline will be substituted for both Hydrogen and Minocycline for intravenous administration. Water will be substituted for hydrogen when administered p.o., and placebo capsules will be substituted for minocycline.
  Placebo Hydrogen: Normal saline solution will be administered intravenously, in place of hydrogen solution.
  Placebo tablets will be dissolved into water for the patient to drink, as the patient's condition permits. This will be administered TID for 3 days.
  Placebo Minocycline: Normal saline solution or placebo capsule will be administered i.v. or p.o. respectively, in place of minocycline.
Period: Treatment Period
Arm/Group | Hydrogen/Minocycline | Placebo Hydrogen/Placebo Minocycline
Started | 6 | 8
Completed | 5 | 8
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Day 45 Follow up
Arm/Group | Hydrogen/Minocycline | Placebo Hydrogen/Placebo Minocycline
Started | 5 | 8
Completed | 5 | 8
Not Completed | 0 | 0
Period: Day 90 Follow up
Arm/Group | Hydrogen/Minocycline | Placebo Hydrogen/Placebo Minocycline
Started | 5 | 8
Completed | 5 | 7
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrogen/Minocycline | Placebo Hydrogen/Placebo Minocycline | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.17 (12.32) | 65.13 (13.92) | 69.00 (13.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 14
NIH Stroke Scale (NIHSS) [Median (Inter-Quartile Range); unit: units on a scale] — 15-item neurologic examination scale for severity of stroke. Ratings for each item are scored with 3 to 5 grades. A total NIHSS of 0 is normal; 1-4 is considered a minor stroke; 5-15 moderate; 16-20 moderate to severe; and 21-42 severe.
  units on a scale | 8.5 [7 to 12] | 12.5 [9 to 19.5] | 9.5 [8 to 18]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Favorable Outcome on the Simplified Modified Rankin Scale (sMRSq)
Description: rating scale to assess level of functional independence for patients post-stroke. Scores range from 0 (no symptoms) to 6 (dead).
  mRS scores at 90 days will be classified as favorable or unfavorable based on the baseline NIHSS measured at time of enrollment. Subjects in the lowest baseline severity tertile (NIHSS 5-7) will need to have a 90 day mRS score of 0 to be considered to have a favorable outcome. Subjects with baseline NIHSS 8-14 will need a 90 day mRS score 0-1 to be considered to have a favorable outcome; those with baseline NIHSS 15-25 will need a 90 day mRS score 0-2 to be considered to have a favorable outcome.
Time Frame: 90 days
Population: Subjects lost to follow are considered to have an unfavorable outcome.
Measure: Number; unit: participants
Arm/Group | Hydrogen/Minocycline | Placebo Hydrogen/Placebo Minocycline
Number analyzed (Participants) | 6 | 8
participants
  Unfavorable outcome | 5 | 7
  Favorable outcome | 1 | 1

2. Secondary Outcome: Simplified Modified Rankin Scale (sMRSq)
Description: rating scale to assess level of functional independence for patients post-stroke. Scores range from 0 (no symptoms) to 6 (dead).
Time Frame: 45 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hydrogen/Minocycline | Placebo Hydrogen/Placebo Minocycline
Number analyzed (Participants) | 5 | 8
score on a scale | 2.8 (1.6) | 3.4 (1.3)

3. Secondary Outcome: NIH Stroke Scale (NIHSS)
Description: 15-item neurologic examination scale for severity of stroke. Ratings for each item are scored with 3 to 5 grades. A total NIHSS of 0 is normal; 1-4 is considered a minor stroke; 5-15 moderate; 16-20 moderate to severe; and 21-42 severe.
Time Frame: 90 days
Population: Per protocol the 90 day follow up is done either in person or by phone. The NIHSS is administered subjects who are able to be seen in-person for the follow-up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hydrogen/Minocycline | Placebo Hydrogen/Placebo Minocycline
Number analyzed (Participants) | 2 | 2
score on a scale | 4 (4.2) | 7.5 (3.5)

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Hydrogen/Minocycline | Placebo Hydrogen/Placebo Minocycline
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/8
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/8
Other Adverse Events (participants affected / at risk) | 5/6 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrogen/Minocycline (N=6) | Placebo Hydrogen/Placebo Minocycline (N=8)
stroke (Cardiac disorders) | 1 (1) | 0 (0)
bradycardia and syncope (Cardiac disorders) | 1 (2) | 0 (0)
hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
thrombus (Cardiac disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrogen/Minocycline (N=6) | Placebo Hydrogen/Placebo Minocycline (N=8)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Hypotension (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
vaginal bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
ecchymotic penis and scrotum (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
hypotension (Cardiac disorders) | 1 (1) | 1 (2)
twitching with anisocoria (Eye disorders) | 0 (0) | 1 (1)
Wound complication (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
skin redness and swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
petechial hemorrhagic stroke conversion (Cardiac disorders) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 1 (1)
inflammation in foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
black lesion in foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
hyponatremia (Renal and urinary disorders) | 1 (1) | 0 (0)
increased BUN/creatinine (Renal and urinary disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
nausea (General disorders) | 0 (0) | 1 (1)
decreased sensation (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT03320018/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT03320018/ICF_001.pdf